CLINICAL TRIAL: NCT07349732
Title: Comparative Study Between Ligamentum Teres Cardiopexy and Gastric Bypass in Treatment of Post Sleeve Gastrectomy GERD
Brief Title: Ligamentum Teres Cardiopexy in Treatment of GERD After Sleeve Gastrectomy
Acronym: GERD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew Mokbel (Other)
Responsible Party: Sponsor-Investigator, Andrew Mokbel, director, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ligamentum teres cardiopexy
Record Dates: First submitted 2025-12-30; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Effect of Ligamentum Teres in Hiatus Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ligamentum teres cardiopexy (Other): will do ligamentum teres cardiopexy in treatment of GERD
  Interventions: Procedure: ligamentum teres cardiopexy

INTERVENTIONS:
Procedure: ligamentum teres cardiopexy — ligamentum ters cardiopexy in tratment of GERD in post sleeve gastrectomy

SUMMARY:
The aim of this study is to evaluate the effectiveness and safety of surgical repair techniques with ligamentum teres cardiopexy on symptomatic relief of gastroesophageal reflux disease (GERD), recurrence rates of hiatus hernia, and overall patient quality of life following sleeve gastrectomy

DETAILED DESCRIPTION:
Laparoscopic sleeve gastrectomy (LSG) has become one of the most commonly performed bariatric procedures worldwide due to its effectiveness in achieving sustained weight loss and improving obesity-related comorbidities. However, it is increasingly recognized that LSG may lead to or exacerbate gastroesophageal reflux disease (GERD) and contribute to the development or worsening of hiatus hernia (HH). GERD incidence after LSG has been reported to range from 20% to 60%, making it a significant postoperative complication impacting patient quality of life. The underlying pathophysiology involves changes in gastroesophageal anatomy and physiology following the resection of the gastric fundus and alteration of the lower esophageal sphincter pressure, along with increased intragastric pressure due to the sleeve's tubular shape Changes after a sleeve gastrectomy

1. Sectioning the gastric fundus leaves the upper esophagus open when the food passes and changes the angle of His from 36° to 51
2. Damaging the sling fibers, cutting the noose that forms the LES, and promoting GERD
3. Augmented intragastric pressure, confirmed by manometry, increases the gastroesophageal pressure gradient and reflux
4. Herniation of the gastric tube into the thoracic cavity, disarming the associated gastro and esophagus-phrenic ligaments, leaving the pouch with a greater capacity to suffer from the pressures applied by the stomach and thorax, which may produce a hiatal hernia (HH)
5. Vagal nerve injury
6. Poor surgical technique leads to twisting, kinking, or strictures of the gastric tube.
7. A dynamic pylorus When Surgery Is Considered

After SG, most patients with GERD are first managed with lifestyle changes and medical therapy (e.g. PPIs). Surgery or more invasive interventions are considered when:

1. GERD symptoms are refractory despite maximal medical treatment.
2. There are anatomical problems contributing to reflux, e.g. hiatal hernia, sleeve twist, stenosis, sleeve dilation, intrathoracic migration of the sleeve.
3. There's also insufficient weight loss or weight regain (so revisional surgery may serve dual purposes).

ELIGIBILITY:
Inclusion Criteria:

* • patients who previously underwent laparoscopic sleeve gastrectomy

  * Adequate anatomy to perform the procedure For example, ability to mobilize adequate intra-abdominal esophagus (e.g. freeing 3-5 cm of esophagus into abdomen) and enough ligamentum teres tissue to wrap/fix
  * Patients experiencing GERD symptoms refractory to medical therapy (e.g., proton pump inhibitors more than 8 weeks )

Exclusion Criteria:

* • Known esophageal motility disorders (achalasia, scleroderma).

  * Barrett's esophagus with high grade dysplasia
  * Presence of complications contraindicating the use of ligamentum teres For example, prior surgeries that compromised ligamentum teres, hepatic disease, malignancy near ligament region

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in GERD symptoms at 6-month and 12-month follow-up. | 12 month
  Development and evaluation of FSSG: frequency scale for the symptoms of GERD

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No